CLINICAL TRIAL: NCT03764189
Title: Evaluation of Micro-osteoperforation on Rate of Maxillary En-masse Retraction: A Randomized Controlled Trial
Brief Title: Evaluation of Micro-osteoperforation on Rate of Maxillary En-masse Retraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nashwa abdel mohsen mohamed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-11-41
Record Dates: First submitted 2018-12-01; First posted 2018-12-05 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Class II Division 1 Malocclusion
Keywords: Accelerated tooth movement AND anterior segment retraction AND miniscrews AND microosteoperforation
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Masking Description: not possible as the subject will sign an informed consent and areas of microosteoperforation will be apparent
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- en masse retraction only (No Intervention): anterior segment retraction on miniscrews without microosteoperforation
- en masse retraction with alveocentesis (Active Comparator): anterior segment retraction on miniscrews with microosteoperforation
  Interventions: Procedure: microosteoperforation

INTERVENTIONS:
Procedure: microosteoperforation — small holes made using large round bur
  Other Names: accelerated tooth movement; alveocentesis
  Arms: en masse retraction with alveocentesis

SUMMARY:
accelerated anterior teeth retraction with the help of microosteoperforation procedure and miniscrews.

DETAILED DESCRIPTION:
the study contains 2 groups each contains 13 subjects, A control group (anterior segment retraction with the help of miniscrews) and an intervention group ( anterior segment retraction with the help of miniscrews and microosteoperforation)

ELIGIBILITY:
Inclusion Criteria:

* Females with an age ranging between 16-30 years.
* Malocclusion that requires bilateral extraction of the maxillary first premolars and anterior segment retraction; Angle class I mal-occlusion with bi-alveolar dental protrusions or class II division 1.
* Healthy dental and periodontal condition with a good oral hygiene
* Absence of degenerative conditions.
* Full set of permanent dentition.

Exclusion Criteria:

* Medically compromised patients.
* Previous orthodontic treatment
* Patients suffering from any congenital, hereditary or systemic diseases or asymmetries that might have an influence on tooth movement
* Chronic use of any medications affecting orthodontic tooth movement (eg: NSAIDs).
* Active periodontal affection or severe gingival inflammation.

Ages: 16 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 13 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Rate of En-masse retraction | three to six months
  retracting six anterior teeth

SECONDARY OUTCOMES:
Root resorption affecting the six anterior teeth. | three to six months
  Amount of root volume loss analyzed through CBCT software
Tipping affecting the anterior teeth. | three to six months
  Changes in angular measurements calculated through CBCT software
Extrusion of anterior teeth | three to six months
  Linear measurement changes in the clinical height using CBCT

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Kaddah, Phd, Study Director — Cairo u
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
All patients' personal data of the patient will be kept safely and no patient data will be used outside the trial unless approved by the patient.

REFERENCES:
- [Background] McGorray SP, Dolce C, Kramer S, Stewart D, Wheeler TT. A randomized, placebo-controlled clinical trial on the effects of recombinant human relaxin on tooth movement and short-term stability. Am J Orthod Dentofacial Orthop. 2012 Feb;141(2):196-203. doi: 10.1016/j.ajodo.2011.07.024. PMID 22284287
- [Background] Nicozisis, J., Accelerated Orthodontics With Alveocentesis. Princeton Orthodontics. Clin Orthod, 2012. 19: p. 1-4
- [Background] Collins MK, Sinclair PM. The local use of vitamin D to increase the rate of orthodontic tooth movement. Am J Orthod Dentofacial Orthop. 1988 Oct;94(4):278-84. doi: 10.1016/0889-5406(88)90052-2. PMID 3177281
- [Background] Blanco, J., et al., Efecto de la administración sistémica del 1, 25 Dihidrxicolecalciferol sobre la velocidad del movimiento ortodóncico en humanos. Estudio Clínico. Revista Odontos, 2001. 8: p. 13-21
- [Background] Cruz DR, Kohara EK, Ribeiro MS, Wetter NU. Effects of low-intensity laser therapy on the orthodontic movement velocity of human teeth: a preliminary study. Lasers Surg Med. 2004;35(2):117-20. doi: 10.1002/lsm.20076. PMID 15334614
- [Background] Alfawal AMH, Hajeer MY, Ajaj MA, Hamadah O, Brad B. Evaluation of piezocision and laser-assisted flapless corticotomy in the acceleration of canine retraction: a randomized controlled trial. Head Face Med. 2018 Feb 17;14(1):4. doi: 10.1186/s13005-018-0161-9. PMID 29454369
- [Background] Alikhani, M., et al. Micro-osteoperforations: minimally invasive accelerated tooth movement. in Seminars in Orthodontics. 2015. Elsevier
- [Background] Alikhani M, Raptis M, Zoldan B, Sangsuwon C, Lee YB, Alyami B, Corpodian C, Barrera LM, Alansari S, Khoo E, Teixeira C. Effect of micro-osteoperforations on the rate of tooth movement. Am J Orthod Dentofacial Orthop. 2013 Nov;144(5):639-48. doi: 10.1016/j.ajodo.2013.06.017. PMID 24182579
- [Background] Ribeiro GL, Jacob HB. Understanding the basis of space closure in Orthodontics for a more efficient orthodontic treatment. Dental Press J Orthod. 2016 Mar-Apr;21(2):115-25. doi: 10.1590/2177-6709.21.2.115-125.sar. PMID 27275623
- [Result] Kau CH, Kantarci A, Shaughnessy T, Vachiramon A, Santiwong P, de la Fuente A, Skrenes D, Ma D, Brawn P. Photobiomodulation accelerates orthodontic alignment in the early phase of treatment. Prog Orthod. 2013 Sep 19;14:30. doi: 10.1186/2196-1042-14-30. PMID 24326198